CLINICAL TRIAL: NCT01303458
Title: Addressing Low-Income Families' Basic Social Needs at Pediatric Visits: the WE CARE Project
Brief Title: Addressing Low-Income Families' Basic Social Needs at Pediatric Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Arvin Garg, Assistant Professor of Pediatrics, Boston Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 4R00HD056160-02 (NIH); 4R00HD056160-02 (NIH)
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Low Income Families Basic Social Needs
Keywords: community resource; well-child care visit; low-income
MeSH Terms: interventions — 6-bromo-2-naphthyl sulfate; Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention arm (Experimental): Study subjects will receive the Basic Needs Surveillance (BNS) intervention.
  Interventions: Behavioral: Basic Needs Surveillance (BNS) protocol
- Control arm (No Intervention): Study subjects in the control arm will receive the standard of care.

INTERVENTIONS:
Behavioral: Basic Needs Surveillance (BNS) protocol — The BNS intervention will consist of 4 components: 1) WE CARE survey which mothers will fill out in the waiting room prior to their child's WCC visits; 2) Family Resource book containing 1-page information sheets on resources, that providers will have access to in exam rooms; 3) a Community Resource Coordinator who will assist families link to available resources, and update providers; 4) Training Session which will provide a 1 hr overview of the intervention to providers
  Arms: Intervention arm

SUMMARY:
This research project is aimed to address low-income families' basic social needs (housing, food, employment, education, childcare, utilities) within the context of pediatric primary care. This project builds upon the PI's prior study at Hopkins which demonstrated a positive impact of a similar intervention on pediatric residents' screening and referral to community agencies. This study will specifically test whether a further strengthened intervention--Basic Needs Surveillance (BNS) protocol-- can lead to greater maternal enrollment in community resources and receipt of eligible benefits. In addition, we will measure the intervention's impact on maternal well-being, and compliance with well-child care (WCC) visits.

The project will take place at eight community health centers in the Greater Boston Area. The centers will be randomized to either an intervention or control site. Mothers who bring their infant in for a WCC visit from birth to 6 months will be eligible. They will be followed until their child is one year of age. Study subjects will complete two self-administered surveys (baseline, follow-up), and one brief telephone interview (when their infant is 9 months old). Pediatric providers will also be subjects; and will fill out a demographic questionnaire at the time of enrollment.

The BNS intervention will consist of 4 components: 1) WE CARE survey which mothers will fill out in the waiting room prior to their child's WCC visits; 2) Family Resource book containing 1-page information sheets on resources, that providers will have access to in exam rooms; 3) a Community Resource Coordinator who will assist families link to available resources, and update providers; 4) Training Session which will provide a 1 hr overview of the intervention to providers.

Families attending the control health centers will receive standard of care. Enrolled mothers will be offered the intervention at the end of the 12-month follow-up interview. When follow-up data collection is complete, the PI will offer the control sites the opportunity to implement the BNS protocol.

ELIGIBILITY:
Inclusion Criteria:

* Mothers (18 yrs or older) who bring their infant between the ages of birth and 6 months for a well-child care visit
* Medical providers who provide care to pediatric patients at the participating community health centers

Exclusion Criteria:

* Foster parent
* Mothers who anticipate changing their infant's site for care
* Mothers who are non-English or non-Spanish speaking
* Infants with hx of prematurity (born before 32 weeks)
* Infants with chronic cardiac or respiratory diseases
* Previously enrolled mother

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Enrollment in new community-based resources and services | when index child is 1 yr of age

SECONDARY OUTCOMES:
Food insecurity | when index child is one yr of age
Maternal depression | when index child is one yr of age
preventative care adherence, child health, child maltreatment | when index child is one yr of age
referrals received by mother at index well-child care visit | 1st well-child care visit
  referrals received for any of the 6 following unmet needs (food, housing, employment, education, childcare, heat)
contact of community resource | child is 9 months of age
  self-report of contact of a community resource for one of the 6 unmet needs (food, housing, employment, childcare, education, heat)
unmet basic needs | 12 month follow-up
  food, housing, employment, education, childcare, heat
parenting stress, maternal life satisfaction | 12 month follow-up

OTHER OUTCOMES:
unmet basic needs | at enrollment
  Questions from Children's HealthWatch survey used to measure 6 needs: food insecurity (18-item US food security scale), housing instability, education i.e., not completed high school, childcare, heat, employment.

CONTACTS AND LOCATIONS:
Overall Officials: Arvin Garg, MD, MPH, Principal Investigator — Boston Medical Center
Locations (9):
- United States (9):
  - Arvin Garg, Boston, Massachusetts
  - Harvard Street Neighborhood Health Center, Dorchester, Massachusetts
  - Dorchester House Multi-Service Center, Dorchester, Massachusetts
  - Neponset Health Center, Dorchester, Massachusetts
  - Codman Square Health Center, Dorchester, Massachusetts
  - Upham's Corner Health Center, Dorchester, Massachusetts
  - Greater Roslindale Medical and Dental Center, Roslindale, Massachusetts
  - The Dimock Center, Roxbury, Massachusetts
  - South Boston Community Health Center, South Boston, Massachusetts

REFERENCES:
- [Derived] Garg A, Toy S, Tripodis Y, Silverstein M, Freeman E. Addressing social determinants of health at well child care visits: a cluster RCT. Pediatrics. 2015 Feb;135(2):e296-304. doi: 10.1542/peds.2014-2888. Epub 2015 Jan 5. PMID 25560448